CLINICAL TRIAL: NCT07311538
Title: A Phase IIa Study to Investigate the Efficacy and Safety of BRY812 for Injection in Patients With LIV-1 Positive Advanced Gynecologic Malignancies
Brief Title: Phase IIa Study of BRY812 Monotherapy in Advanced Gynecological Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRY812-201
Record Dates: First submitted 2025-11-18; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Advanced Gynecological Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (1):
- BRY812 (Experimental)
  Interventions: Drug: BRY812 for injection

INTERVENTIONS:
Drug: BRY812 for injection — BRY812 for injection will be administered by intravenous drip, tentatively once per cycle spanning 3 weeks on D1 of each cycle until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation or withdrawal from the study. The dose of each administration will be calculated based on the weight measured prior to such administration. The dosing regimen (dosing frequency and interval) for subsequent study may be adjusted based on prior data. The intravenous drip should last for ≥ 90 min for the first dose and may be adjusted to ≥ 30 min for subsequent doses if the first dose is tolerable.

SUMMARY:
This study is a single-arm, open-label, multicenter Phase IIa trial designed to evaluate the efficacy, safety, and pharmacokinetic profile of BRY812 for Injection in patients with LIV-1-positive advanced gynecological malignancies. The study comprises two cohorts. For Cohort 1 (ovarian cancer), a Simon's two-stage design is adopted. In the first stage, 13 evaluable subjects will be enrolled. If fewer than 3 subjects achieve an objective response among these 13, enrollment in this cohort will be terminated. Otherwise, the cohort will proceed to the second stage, and additional 23 evaluable subjects will be enrolled, bringing the total to 36. If at least 10 out of the 36 evaluable subjects achieve an objective response, the cohort will be considered worthy of further investigation. Cohort 2 (endometrial cancer and ovarian clear cell carcinoma) plans to enroll approximately 20 subjects in a single stage.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects who voluntarily sign the informed consent form, understand the nature, objectives, and procedure of the study and are able to complete the study according to the protocol;
* (2) Female patients, ≥ 18 years of age (based on the date of signing the informed consent form);
* (3) LIV-1 positive, as assessed by a central laboratory
* (4) Patients with histologically or cytologically confirmed locally advanced or metastatic gynecological malignancies are enrolled into two cohorts:

Cohort 1 (Ovarian Cancer):

Diagnosis of high-grade serous epithelial ovarian cancer (EOC). Must have received 1 to 3 prior lines of systemic anticancer therapy.

Cohort 2 (Endometrial Cancer and Ovarian Clear Cell Carcinoma):

For Endometrial Cancer: Diagnosis of recurrent or metastatic advanced endometrial carcinoma (all histologies except sarcoma). Patients must have received up to 3 prior lines of systemic therapy, platinum-based chemotherapy and anti-PD-1/PD-L1 therapy .

For Ovarian Clear Cell Carcinoma: Pathologically confirmed ovarian clear cell carcinoma. The definitions for prior therapy lines (1-3 lines) are the same as for Cohort 1.

* (5) According to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors), there is at least 1 measurable lesion;
* (6) Radiographic disease progression must have occurred during or after the most recent anti-tumor therapy.
* (7) Eastern Cooperative Oncology Group (ECOG) Status 0 to 1;
* (8) Adequate organ and bone marrow function (no treatment with cells, growth factors, or transfusions within 14 days prior to the first administration), as defined below:

  1. Hematology: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 90 g/L;
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN;
  3. Renal function: creatinine clearance (CrCL) (based on Cockcroft-Gault equation) ≥ 60 mL/min;
* (9) Expected survival ≥ 12 weeks;
* (10) Female subjects with fertility potential must test negative for serum human chorionic gonadotropin (HCG) before they are enrolled in the study. Female subjects with fertility potential or male subjects who have a female partner must agree to maintain no pregnancy plan and take effective contraceptive measures such as condoms from the signing of ICF to 6 months after the last dose of study drug (see Annex 1 for details); females are considered fertile from menarche to menopause (at least 12 months without menstruation) unless they are permanently infertile (through hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Exclusion Criteria:

* (1) Subjects who have previous severe hypersensitivity to BRY812 or known hypersensitivity to any component or excipient of the study drug;
* (2) Subjects who have previously received drugs which target LIV-1, or MMAE-containing drugs, including but not limited to antibody-drug conjugates (ADCs) that utilize MMAE as the cytotoxic payload;
* (3) Subjects who have any active infection requiring systemic therapy by intravenous infusion within 2 weeks prior to the first dose of study drug;
* (4) Subjects who have previous or current presence of two or more primary tumors (excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin, and other tumors that have been stable for more than 5 years after treatment);
* (5) Subjects who have symptoms of active central nervous system metastases, except those with brain parenchymal metastases assessed as stable by the investigator based on the following conditions:

  1. No seizures within > 12 consecutive weeks with or without the treatment of antiepileptic drugs;
  2. Glucocorticoids are not required within the 2 weeks prior to the first dose;
  3. Two consecutive MRI scans (at least 4 weeks apart) show a stable state on imaging;
  4. The conditions remain stable and asymptomatic for more than 1 month after treatment;
* (6) Subjects with serious cardiovascular and cerebrovascular diseases and lung diseases, including but not limited to:

  1. Stroke, intracranial hemorrhage, unstable angina pectoris, congestive heart failure (NYHA class III-IV), myocardial infarction, severe arrhythmias (such as sustained ventricular tachycardia and ventricular fibrillation), congenital long QT syndrome, torsade de pointes, and symptomatic pulmonary embolism within 6 months before enrollment;
  2. Uncontrolled hypertension (at least 2 consecutive measurements of systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
  3. Echocardiogram (ECHO) or multigated acquisition scan (MUGA) shows left ventricular ejection fraction (LVEF) < 50%;
  4. During the screening period, the mean corrected (by Fridercia's formula) QT interval on three consecutive electrocardiograms is prolonged (> 470 ms);
  5. Subjects who have interstitial lung diseases, severe impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, and other lung diseases assessed by the investigator as clinically significant;
* (7) Subjects who have active gastrointestinal bleeding or severe intestinal obstruction;
* (8) Subjects who have undergone major surgery within 4 weeks prior to the first dose of study drug or are expected to be performed during the study;
* (9) Subjects who have a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* (10) Thromboembolic events diagnosed within 6 months prior to the first dose that require therapeutic anticoagulation (except for stable, long-term maintenance anticoagulation for events diagnosed >6 months ago), or known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders). Prophylactic anticoagulation at low doses (e.g., low molecular weight heparin, direct thrombin inhibitors, or factor Xa inhibitors) is permitted;
* (11) Subjects who have used strong inhibitors or substrates of CYP3A4 and/or P-gp within 4 weeks before the first dosing or within 5 half-lives of the used drug (whichever is shorter), or who have received anti-tumor therapy or participated in other clinical studies and used other study drugs, including chemotherapy, targeted therapy, immunotherapy, biotherapy (tumor vaccines, cytokines, or growth factors for cancer control), etc.; or who have received prepared slices of Chinese crude drugs or Chinese patent medicines as anti-tumor treatment within 1 week before the first dose of study drug;
* (12) Subjects who have received radiotherapy within 4 weeks prior to the first dose of the study drug, with specific timelines as follows: within 4 weeks for palliative stereotactic radiotherapy to the abdomen or for whole-brain radiotherapy (WBRT) / wide-field radiotherapy; within 2 weeks for palliative stereotactic radiotherapy to non-abdominal sites or limited-field radiotherapy for symptom relief. Additionally, patients with a history of radiotherapy involving >30% of the bone marrow are excluded.
* (13) Toxicity of previous antineoplastic therapy does not resolve to grade ≤ 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic abnormal laboratory findings considered by the investigator, such as elevated ALP, hyperuricemia, elevated blood glucose, etc.; except for toxicity with no safety risk determined by the investigator, such as alopecia, pigmentation, etc.);
* (14)Subjects with active or chronic corneal disorders, a history of corneal transplantation, or active ocular diseases requiring ongoing treatment/monitoring.
* (15) Subjects who have been vaccinated with a live vaccine within 4 weeks before the first dose, or who intend to be vaccinated with a live vaccine during the study;
* (16) Subjects who have received more than 1 week of treatment with systemic corticosteroids (methylprednisolone > 10 mg/day or an equivalent dose of other similar drug) within 2 weeks prior to the first dose of study drug;
* (17) Subjects who have used immunosuppressants within 2 weeks prior to the first dose or once had active autoimmune diseases or had a prior history of autoimmune diseases;
* (18) Subjects who test positive for Hepatitis B surface antigen (HBsAg) with HBV DNA beyond the normal range; or subjects who test positive for hepatitis B core antibody with HBV DNA beyond the upper limit of normal, but do not agree to regular DNA testing during treatment and follow-up, or do not agree to receive antiviral therapy; subjects who test positive for hepatitis C virus (HCV) antibody and HCV RNA; subjects who are seropositive for human immunodeficiency virus (HIV); subjects who have syphilis and need to receive systemic treatment;
* (19) Subjects who have any mental or cognitive disorders that may limit their understanding and execution of the informed consent form;
* (20) Subjects who are pregnant or breastfeeding;
* (21) Subjects who are not eligible for enrollment or may not be able to complete the study due to other reasons by the investigator's assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessment (RECIST v1.1) | Baseline, every 6 weeks after first dose up to 24 weeks, every 12 weeks thereafter, through study completion, an average of 6 months
  The Objective Response Rate (ORR) and other efficacy outcomes will be evaluated by an Independent Review Committee (IRC) using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Safety assessment (NCI CTCAE v5.0) | Immediately after the intervention, through study completion, an average of 6 months
  Safety assessments: NCI CTCAE v5.0 is mainly used to evaluate safety indicators include physical examination, vital signs, laboratory tests, 12-lead electrocardiogram, other safety-related tests, and AEs.
Pharmacokinetic assessment | Immediately after the intervention, through study completion, an average of 6 months
  The concentrations of BRY812, total antibody and free monomethyl auristatin E (MMAE) in blood will be determined, and the following parameters will be calculated respectively.
Immunogenicity assessment | Immediately after the intervention, through study completion, an average of 6 months
  The anti-drug antibody (ADA) of BRY812 in the blood is detected, and the antibody titer of ADA-positive patients is further detected according to the situation, and whether they have neutralizing antibody (NAb) is detected if necessary.

IPD SHARING:
Plan to Share IPD: No